CLINICAL TRIAL: NCT00262067
Title: A Multicenter, Phase III, Randomized, Placebo-controlled Trial Evaluating the Efficacy and Safety of Bevacizumab in Combination With Chemotherapy Regimens in Subjects With Previously Untreated Metastatic Breast Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Bevacizumab in Combination With Chemotherapy in Untreated Metastatic Breast Cancer (RIBBON 1)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF3694g; BO20094 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Results first posted 2013-10-25 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bevacizumab + chemotherapy (Experimental): Patients received bevacizumab 15 mg/kg intravenously (IV) on Day 1 of every 21-day cycle plus one of several standard chemotherapies (taxanes, anthracycline-based regimens, or capecitabine) for metastatic breast cancer.
  Interventions: Drug: Bevacizumab; Drug: Chemotherapy
- Placebo + chemotherapy (Placebo Comparator): Patients received placebo to bevacizumab administered IV on Day 1 of every 21-day cycle + 1 of several standard chemotherapies (taxanes, anthracycline-based regimens, or capecitabine) for metastatic breast cancer.
  Interventions: Drug: Placebo; Drug: Chemotherapy

INTERVENTIONS:
Drug: Bevacizumab — Patients received bevacizumab until disease progression, treatment limiting toxicity, or death due to any cause up to a maximum treatment duration of 48 months. The dose of bevacizumab was based on the patient's weight at either screening or baseline and remained the same throughout the blinded treatment phase of the study. The initial dose was delivered over 90±10 minutes. If there were no infusion related adverse events (fever and/or chills), the second infusion was delivered over 60±10 minutes. If the 60 minute infusion was well tolerated, all subsequent infusions were delivered over 30±10 minutes.
  Other Names: Avastin
  Arms: Bevacizumab + chemotherapy
Drug: Placebo — Placebo consisted of the vehicle for bevacizumab without the antibody.
  Arms: Placebo + chemotherapy
Drug: Chemotherapy — The chemotherapy was selected by the investigator prior to randomization. Chemotherapy treatment continued until disease progression, unacceptable toxicity, investigator/patient decision, or death, whichever occurred first, except for the anthracycline-based regimens, which had a maximum treatment duration of 8 cycles.
  Taxanes - 1 of the following 2 taxanes on Day 1 of every 21-day cycle
  1. Docetaxel 75-100 mg/m^2 IV
  2. Paclitaxel protein-bound particles (Abraxane®) 260 mg/m^2 IV
  Anthracyclines - 1 of the following 4 anthracycline-based regimens on Day 1 of every 21-day cycle
  1. 5-fluorouracil 500 mg/m^2 IV + epirubicin 90-100 mg/m^2 IV + cyclophosphamide 500 mg/m^2 IV
  2. 5-fluorouracil 500 mg/m^2 IV + doxorubicin 50 mg/m^2 IV + cyclophosphamide 500 mg/m^2 IV
  3. Doxorubicin 50-60 mg/m^2 IV + cyclophosphamide 500-600 mg/m^2 IV
  4. Epirubicin 90-100 mg/m^2 IV + cyclophosphamide 500-600 mg/m^2 IV
  Capecitabine: 1000 mg/m^2 orally twice daily on Days 1-14 of each 21-day cycle

SUMMARY:
This is a Phase III, multicenter, randomized, placebo-controlled trial designed to evaluate the efficacy and safety of bevacizumab in combination with chemotherapy compared with chemotherapy alone in subjects with previously untreated metastatic breast cancer.

DETAILED DESCRIPTION:
This study includes a blinded treatment phase, an optional open-label post-progression phase, and a survival follow-up phase. During the blinded treatment phase, patients receive chemotherapy and study drug (bevacizumab or placebo) every 3 weeks until disease progression, treatment-limiting toxicity, or death due to any cause. The optional open-label post-progression phase consists of chemotherapy treatment (per investigator discretion) and optional treatment with open-label bevacizumab. Patients who complete the study or who discontinue from treatment (regardless of participation in the optional open-label post-progression phase) will be followed for survival and subsequent anti-cancer therapies every 4 months until death, withdrawal of consent, loss to follow-up, or study termination. Patients who discontinue from treatment during the blinded treatment phase for reasons other than disease progression will have tumor assessments every 9 weeks until documented disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast, with measurable or non-measurable locally recurrent or metastatic disease.
* Signed Informed Consent Form.
* Age ≥ 18 years.
* For women of childbearing potential, use of accepted and effective method of non-hormonal contraception.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Ability and capacity to comply with study and follow-up procedures.
* For anthracycline cohort only: Adequate left ventricular function at study entry, defined as a left ventricular ejection fraction (LVEF) ≥ 50% by either multigated acquisition (MUGA) scan scan or echocardiography (ECHO).
* For subjects who have received recent radiation therapy, recovery prior to baseline (Day 0) from any significant (Grade ≥ 3) acute toxicity.

Exclusion Criteria:

* Unknown human epidermal growth factor receptor 2 (HER2) status or known HER2-positive status.
* Prior chemotherapy for locally recurrent or metastatic disease.
* Prior hormonal therapy less than 1 week prior to Day 0.
* Prior adjuvant or neoadjuvant chemotherapy within 12 months prior to Day 0.
* For anthracycline cohort only: Prior anthracycline as part of neoadjuvant or adjuvant therapy for localized breast cancer.
* Investigational therapy within 28 days of Day 0.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures, such as fine needle aspirations or core biopsies, within 7 days prior to Day 0.
* Prior therapy with bevacizumab, sorafenib, sunitinib, or other vascular endothelial growth factor (VEGF) pathway-targeted therapy.
* Known brain or other central nervous system (CNS) metastases.
* Blood pressure of > 150/100 mmHg.
* Unstable angina.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF).
* History of myocardial infarction within 6 months prior to Day 0.
* History of stroke or transient ischemic attack within 6 months prior to Day 0.
* Clinically significant peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0.
* Serious non-healing wound, ulcer, or bone fracture.
* Pregnancy (positive serum pregnancy test) or lactation.
* Inadequate organ function, as evidenced by any of the following laboratory values: Absolute neutrophil count < 1500/uL; platelet count < 100,000/uL; total bilirubin > 1.5 mg/dL; alkaline phosphatase, AST, and/or ALT > 2x upper limit of normal (ULN) (> 5x ULN in subjects with known liver or, for alkaline phosphatase elevations, bone involvement); alkaline phosphatase > 2x ULN (> 7x ULN in subjects with known bone involvement); serum creatinine > 2.0 mg/dL; partial thromboplastin time (PTT) and/or either international normalized ratio (INR) or prothrombin time (PT) > 1.5x upper limit of normal (except for subjects receiving anti-coagulation therapy); urine protein/creatinine ratio > 1.0 at screening for U.S. subjects, or urine dipstick for proteinuria >/= 1+ at screening followed by 24-hour urine collection demonstrating > 1 g protein/24 hr for ex-U.S. subjects.
* Uncontrolled serious medical or psychiatric illness.
* Active infection requiring intravenous (iv) antibiotics at Day 0.
* History of other malignancies within 5 years of Day 0 except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix (subjects with a history of bilateral breast cancer will be eligible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1237 (Actual)
Dates: Start 2005-12; Primary Completion 2008-07 (Actual); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Faoro, MD, Study Director — Genentech, Inc.
Locations (84):
- United States (5):
  - Fullerton, California
  - Santa Barbara, California
  - Iowa City, Iowa
  - Sioux City, Iowa
  - Wichita, Kansas
- Australia (8):
  - Geelong
  - Malvern
  - Melbourne
  - Perth
  - Southport
  - Wahroonga
  - Waratah
  - Wollongong
- Brazil (5):
  - Porto Alegre
  - Rio de Janeiro
  - Salvador
  - Santo André
  - São Paulo
- Canada (2):
  - Winnipeg, Manitoba
  - Montreal, Quebec
- France (5):
  - Marseille
  - Paris
  - Reims
  - Saint-Herblain
  - Strasbourg
- Greece (5):
  - Athens
  - Chania
  - Heraklion
  - Pátrai
  - Thessaloniki
- Guatemala City, Guatemala
- Mexico (4):
  - Acapulco
  - Aguascalientes
  - Mérida
  - Monterrey
- Netherlands (3):
  - Amstelveen
  - Apeldoorn
  - Delft
- Oslo, Norway
- Panama City, Panama
- Callao, Peru
- Quezon City, Philippines
- Russia (10):
  - Chelyabinsk
  - Ivanovo
  - Kazan'
  - Moscow
  - Novosibirsk
  - Obninsk
  - Ryazan
  - Saint Petersburg
  - Samara
  - Ufa
- Singapore, Singapore
- South Korea (2):
  - Kyunggi-do
  - Seoul
- Spain (10):
  - A Coruña
  - Córdoba
  - Elche
  - Girona
  - Madrid
  - San Cristóbal de La Laguna
  - Santander
  - Seville
  - Valencia
  - Zaragoza
- Sweden (3):
  - Gävle
  - Örebro
  - Uppsala
- Taiwan (2):
  - Tainan
  - Taoyuan District
- Ukraine (6):
  - Cherkassy
  - Dnipropetrovsk
  - Kiev
  - Lviv
  - Odesa
  - Zaporizhzhya
- United Kingdom (7):
  - Chelsmford
  - Cottingham
  - Epping
  - Huddersfield
  - Nottingham
  - Sheffield
  - Swansea
- Montevideo, Uruguay

REFERENCES:
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen: Patients received bevacizumab 15 mg/kg intravenously (IV) on Day 1 of every 21-day cycle + either a taxane or anthracycline-based standard chemotherapy for metastatic breast cancer.
- Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen: Patients received placebo to bevacizumab administered IV on Day 1 of every 21-day cycle + either a taxane or anthracycline-based standard chemotherapy for metastatic breast cancer.
- Bevacizumab 15 mg/kg + Capecitabine: Patients received bevacizumab 15 mg/kg intravenously (IV) on Day 1 of every 21-day cycle + capecitabine standard chemotherapy for metastatic breast cancer.
- Placebo to Bevacizumab + Capecitabine: Patients received placebo to bevacizumab administered IV on Day 1 of every 21-day cycle + capecitabine standard chemotherapy for metastatic breast cancer.
Period: Overall Study
Arm/Group | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen | Bevacizumab 15 mg/kg + Capecitabine | Placebo to Bevacizumab + Capecitabine
Started | 415 | 207 | 409 | 206
Completed | 196 | 107 | 193 | 93
Not Completed | 219 | 100 | 216 | 113
Not completed — Death | 190 | 89 | 186 | 99
Not completed — Lost to Follow-up | 5 | 4 | 7 | 5
Not completed — Sponsor's Decision to Terminate Study | 1 | 0 | 0 | 0
Not completed — Patient Withdrew for Survival Follow-up | 23 | 7 | 23 | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized patients, regardless of whether they received any study drug or completed the full course of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen | Bevacizumab 15 mg/kg + Capecitabine | Placebo to Bevacizumab + Capecitabine | Total
Number analyzed (Participants) | 415 | 207 | 409 | 206 | 1237
Age, Customized [Number; unit: Participants]
  < 40 years | 29 | 14 | 21 | 15 | 79
  40-64 years | 295 | 160 | 289 | 137 | 881
  ≥ 65 years | 91 | 33 | 99 | 54 | 277
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 413 | 207 | 408 | 204 | 1232
  Male | 2 | 0 | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: PFS was defined as the time from randomization to first documented disease progression (PD) as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) or death due to any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Target lesions should be selected on the basis of their size (those with the longest diameter) and their suitability for accurate repeated measurements by imaging techniques or clinically. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions.
Time Frame: Baseline to the data cut-off date of 31 Jul 2008 (up to 2 years, 7 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen | Bevacizumab 15 mg/kg + Capecitabine | Placebo to Bevacizumab + Capecitabine
Number analyzed (Participants) | 415 | 207 | 409 | 206
Months | 9.2 [8.6 to 10.1] | 8.0 [6.7 to 8.4] | 8.6 [8.1 to 9.5] | 5.7 [4.3 to 6.2]

2. Secondary Outcome: Objective Response as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: An objective response was defined as a complete response or a partial response determined on two consecutive occasions ≥ 4 weeks apart as determined by the investigator using RECIST. For target lesions, a complete response was defined as the disappearance of all target lesions; a partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. For non-target lesions, a complete response was defined as the disappearance of all non-target lesions; a partial response was defined as the persistence of 1 or more non-target lesions.
Time Frame: Baseline to the data cut-off date of 31 Jul 2008 (up to 2 years, 7 months)
Population: Intent-to-treat population: All randomized patients, regardless of whether they received any study drug or completed the full course of treatment. Only patients with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen | Bevacizumab 15 mg/kg + Capecitabine | Placebo to Bevacizumab + Capecitabine
Number analyzed (Participants) | 345 | 177 | 325 | 161
Percentage of participants | 51.3 [45.9 to 56.7] | 37.9 [30.7 to 45.2] | 35.4 [30.2 to 40.6] | 23.6 [17.6 to 30.7]

3. Secondary Outcome: Duration of Objective Response as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Duration of objective response was defined as the time from the first tumor assessment that led to a determination of an objective response to the time of disease progression or death due to any cause, whichever occurred first.
Time Frame: Baseline to the data cut-off date of 31 Jul 2008 (up to 2 years, 7 months)
Population: Intent-to-treat population: All randomized patients, regardless of whether they received any study drug or completed the full course of treatment. Only patients with measurable disease at baseline and who had an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen | Bevacizumab 15 mg/kg + Capecitabine | Placebo to Bevacizumab + Capecitabine
Number analyzed (Participants) | 177 | 67 | 115 | 38
Months | 8.3 [7.2 to 10.7] | 7.1 [6.2 to 8.8] | 9.2 [8.5 to 10.4] | 7.2 [5.1 to 9.3]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause.
Time Frame: Baseline to the data cut-off of 23 Feb 2009 (up to 3 years, 2 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen | Bevacizumab 15 mg/kg + Capecitabine | Placebo to Bevacizumab + Capecitabine
Number analyzed (Participants) | 415 | 207 | 409 | 206
Months | 27.5 [25.6 to 31.4] | NA [23.6 to NA] — The median and the upper limit of the confidence interval could not be estimated due to too few events. | 25.7 [22.0 to 28.4] | 22.8 [20.5 to 28.4]

5. Secondary Outcome: 1-year Survival
Description: 1-year survival was defined as the percentage of patients who were alive 1 year after randomization.
  The percentage of patients alive at 1 year was determined using Kaplan-Meier analyses and the 95% confidence intervals were computed using the Brookmeyer-Crowley method.
Time Frame: Baseline to the data cut-off of 23 Feb 2009 (up to 3 years, 2 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen | Bevacizumab 15 mg/kg + Capecitabine | Placebo to Bevacizumab + Capecitabine
Number analyzed (Participants) | 415 | 207 | 409 | 206
Percentage of participants | 80.7 [76.8 to 84.5] | 83.2 [78.1 to 88.4] | 81.0 [77.1 to 84.8] | 74.8 [68.7 to 80.8]

6. Secondary Outcome: Progression-free Survival (PFS) as Determined by the Independent Review Committee Using Response Evaluation Criteria in Solid Tumors (RECIST)
Description: PFS was defined as the time from randomization to first documented disease progression (PD) as determined by the Independent Review Committee using Response Evaluation Criteria in Solid Tumors (RECIST) or death due to any cause, whichever occurred first.
Time Frame: Baseline to the data cut-off date of 31 Jul 2008 (up to 2 years, 7 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen | Bevacizumab 15 mg/kg + Capecitabine | Placebo to Bevacizumab + Capecitabine
Number analyzed (Participants) | 415 | 207 | 409 | 206
Months | 10.7 [9.9 to 12.1] | 8.3 [8.0 to 9.9] | 9.8 [8.4 to 10.4] | 6.2 [4.7 to 7.8]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the first treatment until 30 days after the last treatment during the blinded treatment phase or the start date of the optional open-label treatment phase, whichever occurred first (up to 3 years 2 months).
Description: Safety population: All randomized patients who received any study treatment, defined as at least 1 full or partial dose of either study drug or chemotherapy. There were a total of 1220 patients in the safety population.
Arm/Group | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen | Bevacizumab 15 mg/kg + Capecitabine | Placebo to Bevacizumab + Capecitabine
Serious Adverse Events (participants affected / at risk) | 156/413 | 59/202 | 140/404 | 72/201
Other Adverse Events (participants affected / at risk) | 91/413 | 19/202 | 72/404 | 15/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen (N=413) | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen (N=202) | Bevacizumab 15 mg/kg + Capecitabine (N=404) | Placebo to Bevacizumab + Capecitabine (N=201)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 3 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 26 | 11 | 3 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 10 | 5 | 3 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 1 | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 7 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 1
Macular hole (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 0 | 6 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 5 | 0 | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ileal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Jejunitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3 | 4 | 3
Asthenia (General disorders) | 2 | 0 | 0 | 2
Chest pain (General disorders) | 3 | 1 | 2 | 3
Death (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 6 | 1
Pain (General disorders) | 3 | 2 | 1 | 1
Pyrexia (General disorders) | 4 | 1 | 7 | 2
Sudden death (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Breast cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 3 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 8 | 1 | 2 | 2
Central line infection (Infections and infestations) | 0 | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 2 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 2
Herpes oesophagitis (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 4 | 1 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 5 | 6 | 5
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0
Salpingo-oophoritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 6 | 1 | 4 | 3
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Sweat gland infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Renal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood potassiumiIncreased (Investigations) | 0 | 1 | 0 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 0
Rotavirus test positive (Investigations) | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 1 | 6 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid sinus syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Coma hepatic (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 2 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 2 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 3 | 1 | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 3 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 1 | 3 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 1 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 7 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 7 | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 9 | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 1 | 3 | 2
Hypertension (Vascular disorders) | 5 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 15 mg/kg + Taxane or Anthracycline-based Regimen (N=413) | Placebo to Bevacizumab + Taxane or Anthracycline-based Regimen (N=202) | Bevacizumab 15 mg/kg + Capecitabine (N=404) | Placebo to Bevacizumab + Capecitabine (N=201)
Neutropenia (Blood and lymphatic system disorders) | 21 | 4 | 16 | 5
Left ventricular dysfunction (Cardiac disorders) | 21 | 8 | 3 | 2
Proteinuria (Renal and urinary disorders) | 22 | 1 | 13 | 0
Hypertension (Vascular disorders) | 39 | 8 | 50 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.